CLINICAL TRIAL: NCT00960284
Title: Randomized Phase II-III Trial of Post-operative Treatment of Pancreatic Adenocarcinoma: Gemcitabine Versus PEFG Followed by Radiochemotherapy With Concomitant Continuous Infusion of 5-fluorouracil
Brief Title: Gemcitabine or Combination Chemotherapy Followed by Chemoradiation for Stage IB, II, or III Pancreatic Cancer
Acronym: PACT-7
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000641309; PACT-7 (Other: IRCCS San Raffaele)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Pancreatic Cancer
Keywords: stage IB pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Cisplatin; Epirubicin; Fluorouracil; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive gemcitabine hydrochloride IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride
- Arm II (Experimental): Patients receive cisplatin IV over 1 hour and epirubicin hydrochloride IV on day 1 and gemcitabine hydrochloride IV over 1 hour on days 1 and 8. Patients also receive fluorouracil IV continuously beginning on day 1 or oral capecitabine. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: capecitabine — Given orally
  Other Names: XELODA
  Arms: Arm II
Drug: cisplatin — Given IV
  Other Names: Cisplatino-TEVA
  Arms: Arm II
Drug: epirubicin hydrochloride — Given IV
  Other Names: Farmarubicina
  Arms: Arm II
Drug: fluorouracil — Given IV
  Other Names: FLuorouracile-TEVA
  Arms: Arm II
Drug: gemcitabine hydrochloride — Given IV
  Other Names: Gemzar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride, cisplatin, epirubicin hydrochloride, fluorouracil, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether gemcitabine hydrochloride is more effective when given alone or together with combination chemotherapy and radiation therapy in treating patients with pancreatic cancer.

PURPOSE: This randomized phase II/III trial is studying gemcitabine hydrochloride to see how well it works when given alone or together with combination chemotherapy and radiation therapy in treating patients with stage IB, stage II, or stage III pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the 1-year progression-free survival of patients with stage IB, II, or III adenocarcinoma of the pancreas treated with adjuvant therapy comprising gemcitabine with vs without cisplatin, epirubicin hydrochloride, and fluorouracil followed by chemoradiotherapy with fluorouracil or capecitabine. (Phase II)
* Compare the 2-year overall survival of patients treated with these regimens. (Phase III)

Secondary

* Assess the feasibility and toxicity of these regimens in these patients.
* Assess the impact of these regimens on the quality of life of these patients.
* Assess the pattern of relapse in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center and radical surgery. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive cisplatin IV over 1 hour and epirubicin hydrochloride IV on day 1 and gemcitabine hydrochloride IV over 1 hour on days 1 and 8. Patients also receive fluorouracil IV continuously beginning on day 1 or oral capecitabine. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Beginning 2-4 weeks after the completion of chemotherapy, patients in both arms undergo radiotherapy 5 days a week for 6 weeks. Patients also receive concurrent fluorouracil IV continuously or oral capecitabine during radiotherapy.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Stage IB-III disease
* Has undergone surgery with radical intent (R0 or R1) within the past 2 months

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100% (90-100% for patients 71-75 years of age)
* WBC ≥ 3,500/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 2 mg/dL
* SGOT and SGPT ≤ 2 times upper limit of normal
* Not pregnant or nursing
* No other malignancy within the past 5 years except surgically treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin
* No psychological, familial, sociological, or geographical condition that would potentially hinder study compliance or follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy for pancreatic adenocarcinoma
* No other concurrent experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
1-year progression-free survival (Phase II) | every 3 months during the first 2 years, every 6 months afterwards

SECONDARY OUTCOMES:
Pattern of relapse | every 3 months during the first 2 years, every 6 months afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- Istituto Scientifico H. San Raffaele, Milan, Italy

REFERENCES:
- [Background] Reni M, Passoni P, Bonetto E, Balzano G, Panucci MG, Zerbi A, Ronzoni M, Staudacher C, Villa E, Di Carlo V. Final results of a prospective trial of a PEFG (Cisplatin, Epirubicin, 5-Fluorouracil, Gemcitabine) regimen followed by radiotherapy after curative surgery for pancreatic adenocarcinoma. Oncology. 2005;68(2-3):239-45. doi: 10.1159/000086780. Epub 2005 Jul 7. PMID 16015040